CLINICAL TRIAL: NCT04441541
Title: The Effects of Treadmill With Biofeedback on Gait Symmetry in Individuals With Chronic Stroke
Brief Title: Treadmill With Biofeedback on Gait Symmetry After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM109073F
Record Dates: First submitted 2020-06-14; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Stroke Syndrome
Keywords: Gait training; Biofeedback; Treadmill; Gait symmetry
MeSH Terms: conditions — Stroke | interventions — Feedback, Sensory

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treadmill with auditory feedback group (Experimental)
  Interventions: Other: Treadmill with auditory feedback
- Treadmill with visual feedback group (Experimental)
  Interventions: Other: Treadmill with visual feedback
- Treadmill with auditory and visual feedback group (Experimental)
  Interventions: Other: Treadmill with auditory and visual feedback
- Treadmill training group (Active Comparator)
  Interventions: Other: Treadmill training

INTERVENTIONS:
Other: Treadmill with auditory feedback — Participants will receive training 3 times per week for 4 weeks (12 sessions).
  Arms: Treadmill with auditory feedback group
Other: Treadmill with visual feedback — Participants will receive training 3 times per week for 4 weeks (12 sessions).
  Arms: Treadmill with visual feedback group
Other: Treadmill with auditory and visual feedback — Participants will receive training 3 times per week for 4 weeks (12 sessions).
  Arms: Treadmill with auditory and visual feedback group
Other: Treadmill training — Participants will receive training 3 times per week for 4 weeks (12 sessions).
  Arms: Treadmill training group

SUMMARY:
This study aims to investigate the immediate, accumulated, and maintainable effects of treadmill with biofeedback on gait symmetry in individuals with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Single stroke experience
* Chronic stroke phase: stroke duration ≥ 6 months
* Independent gait: Functional Ambulation Category (FAC) ≥ 3

Exclusion Criteria:

* Cognitive problem (MMSE < 24)
* Visual or audio deficiency that might affect training
* Severe heart insufficiency or uncontrolled arterial hypertension
* Orthopedic disorders that affecting their gait

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Spatial and temporal gait symmetry | Change from baseline at the first day, 4 weeks, and 8 weeks
  Temporal symmetry ratio: 1-(single support time of affected limb/single support time of unaffected limb)

SECONDARY OUTCOMES:
Walking speed | Change from baseline at the first day, 4 weeks, and 8 weeks
6 Minute Walk Test | Change from baseline at the first day, 4 weeks, and 8 weeks
Timed up and Go test | Change from baseline at the first day, 4 weeks, and 8 weeks
Stroke Impact Scale | Change from baseline at the first day, 4 weeks, and 8 weeks
  quality of life